CLINICAL TRIAL: NCT03900247
Title: Restore Motor Function Through Robotic Arm Exoskeleton and Brain Computer Interface
Acronym: REMAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University (Other); The Danish National Rehabilitation Center for Neuromuscular Diseases (Unknown); Bioservo Technologies AB, Sweden (Unknown); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 6153-00010A
Record Dates: First submitted 2019-03-18; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: brain computer interface
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: REMAP EEG based BCI and SEM-Glove BioServo — EEG-based brain computer interface (BCI) will be adapted to individual ALS patients and modified to control external robotic devices

SUMMARY:
The current project will aid patients with motor impairment to reduce the need for homecare. Specifically the aim is to develop and implement a robotic exoskeleton and brain computer interface to assist and eventually perform arm and hand movement in patients with the progressive neurodegenerative disease ALS. This proposal brings together state-of-the-art robotic technology, EEG-based brain computer interface (BCI) know-how, clinical expertise, patient perspective and industrial partners to develop and implement a robotic arm/hand device that will adapt, with increasing brain-computer control, based on the need of the patient. In short the BCI will measure electroencephalography (EEG) from the surface of the scalp and recognize signature EEG as the patient intents to move. As the patient loses muscle power the BCI robotic-device will gradually take over and support motor activity, even when the patient is totally paralyzed. As the device supports hand/arm function only, the investigators aim to address ADLs associated to hand function, specifically eating activities.

ELIGIBILITY:
Inclusion Criteria:

* ALS according to the latest revision of El Escorial Criteria (Ludorph et al. 2015)
* Loss of muscle force or fine motor skills in a hand

Exclusion Criteria:

* Other severe Neurological or Psychiatric disease
* Drug or Alcohol dependency
* Pregnancy
* Severe cognitive disturbances found to impede with study completion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Action Research Armtest part b Grip | At 6 months
  performance with and without BCI/robotic device

SECONDARY OUTCOMES:
Grip strength | At 6 months
  Hand held dynamometer with and without BCI/robotic device
Bringing glass of water to the mouth | At 6 months
  Ability to bring a glass of water to the mouth with and without BCI/robotic device

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Functionally Integrative Neuroscience, Aarhus, Denmark